CLINICAL TRIAL: NCT00004189
Title: A Phase I and Pharmacokinetic Study of Sequences of NSC 655649 (Rebeccamycin Analogue) and Cisplatin Without and With Granulocyte Colony-Stimulating Factor Support Every 21 Days
Brief Title: Rebeccamycin Analog and Cisplatin With or Without Filgrastim in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067430; UTHSC-IDD-98-34; SACI-IDD-98-34; NCI-T98-0069
Record Dates: First submitted 2000-01-21; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2003-09

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; becatecarin; Cisplatin

ARMS (1):
- Arm I (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: becatecarin; Drug: cisplatin

INTERVENTIONS:
Biological: filgrastim
Drug: becatecarin
Drug: cisplatin

SUMMARY:
Phase I trial to study the effectiveness of rebeccamycin analog and cisplatin with or without filgrastim in treating patients who have advanced cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated doses of a rebeccamycin analogue and cisplatin with or without filgrastim (G-CSF) in patients with advanced malignancies.

II. Determine the qualitative and quantitative toxicities of these regimens in these patients.

III. Determine if the pharmacokinetics of a rebeccamycin analogue are affected by cisplatin and if there are sequence dependent pharmacokinetic effects.

IV. Assess any antitumor effects of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study of a rebeccamycin analogue and cisplatin.

Part I (previously untreated or minimally pretreated patients): The first patient of each cohort receives cisplatin IV over 1 hour followed 2 hours later by a rebeccamycin analogue IV over 1 hour on day 1. The second patient in the same cohort receives the same drugs in the reverse order. The drug sequence for each additional patient within the same cohort is alternated with reference to the preceding patient. During each subsequent course, the study drugs are administered to each patient in the reverse order as compared to the prior course. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Dose escalation is initially performed without filgrastim (G-CSF). Cohorts of 4-6 patients receive escalating doses of a rebeccamycin analogue and cisplatin until the maximum tolerated dose (MTD) of each drug is determined. The MTD is defined as the highest dose at which less than 2 of 6 patients experience dose limiting toxicity (DLT). If 2 of the first 6 patients experience DLT, then dose escalation proceeds in combination with G-CSF treatment. Patients receive G-CSF subcutaneously daily beginning on day 2 and continuing until blood counts have recovered for 2 days or until approximately day 15. Cohorts of 4-6 patients receive escalating doses of a rebeccamycin analogue and cisplatin as above. The MTD is defined as above.

Part II (heavily pretreated patients): Heavily pretreated patients receive a rebeccamycin analogue and cisplatin starting at 2 dose levels preceding the MTD from part I.

Patients are followed for at least 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven advanced malignancy that is refractory to prior therapy or unlikely to benefit from standard therapy (e.g., chemotherapy, radiotherapy, and surgery)

  * Part I: Previously untreated OR minimally pretreated

    * Ineligible for part I and considered heavily pretreated if:

      * Prior radiotherapy to wide ports involving the pelvis or at least 25% of bone marrow
      * Greater than 6 courses of prior combination chemotherapy including alkylating agent
      * Prior nitrosoureas or mitomycin
      * Widespread bone metastases with bone marrow involvement by bone marrow biopsy (positive bilateral bone marrow biopsy for lymphoma patients)
  * Part II: Heavily pretreated as defined above
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Hemoglobin greater than 9 mg/dL
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* No uncontrolled hypertension
* No angina pectoris
* No clinically significant, multifocal, uncontrolled cardiac dysrhythmias

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active serious infection
* No clinically severe peripheral neuropathy (grade 1 or worse)
* No nonmalignant medical condition that would preclude compliance or increase risk of participation in study
* No hypersensitivity to E. coli derived drug preparations

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No other concurrent colony stimulating factors for prophylactic purposes

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks since prior nitrosoureas and mitomycin) and recovered

Endocrine therapy:

* No chronic oral corticosteroids
* No concurrent corticosteroids except as prophylactic antiemetic

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Other:

* At least 1 month since prior investigational agent
* No prophylactic oral or IV antibiotics for neutropenia unless fever present
* No other concurrent anticancer treatment or investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1999-10; Primary Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hammond, MD, Study Chair — The University of Texas Health Science Center at San Antonio
Locations (3):
- United States (3):
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - St. Luke's Lutheran Hospital, San Antonio, Texas